CLINICAL TRIAL: NCT01703845
Title: A Randomised, Open-label, Parallel-group Trial to Assess Pharmacokinetics and Safety of Tiotropium + Olodaterol Fixed-dose Combination (2.5 µg/ 5 µg, 5 µg/ 5 µg) Delivered by the RESPIMAT Inhaler After 3 Weeks Once Daily Treatment in Japanese Patients With Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: A Study to Characterize Pharmacokinetics of Tiotropium + Olodaterol Fixed-dose Combination in Japanese Patients With COPD.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1237.24
Record Dates: First submitted 2012-10-08; First posted 2012-10-11 (Estimated); Results first posted 2015-07-15 (Estimated); Last update posted 2015-07-15 (Estimated); Status verified 2015-06

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Tiotropium Bromide; olodaterol

ARMS (2):
- Tiotropium + Olodaterol (high dose) (Experimental): Tiotropium and Olodaterol fixed dose combination (FDC) solution for inhalation - RESPIMAT
  Interventions: Drug: Tiotropium (high dose) + Olodaterol
- Tiotropium + Olodaterol (low dose) (Experimental): Tiotropium and Olodaterol fixed dose combination (FDC) solution for inhalation - RESPIMAT
  Interventions: Drug: Tiotropium (low dose) + Olodaterol

INTERVENTIONS:
Drug: Tiotropium (high dose) + Olodaterol — Tiotropium + Olodaterol solution for inhalation
  Arms: Tiotropium + Olodaterol (high dose)
Drug: Tiotropium (low dose) + Olodaterol — Tiotropium + Olodaterol solution for inhalation
  Arms: Tiotropium + Olodaterol (low dose)

SUMMARY:
The primary objective of this study is to assess pharmacokinetics of tiotropium + olodaterol fixed-dose combination (2.5 µg/ 5 µg, 5 µg/ 5 µg) delivered by the RESPIMAT inhaler after 3 weeks once daily treatment in Japanese patients with COPD.

ELIGIBILITY:
Inclusion criteria:

1. Diagnosis of chronic obstructive pulmonary disease
2. Relatively stable airway obstruction with post FEV1=<30% of predicted normal and< 80% predicted normal and post FEV1/FVC <70%
3. Male or female Japanese patients, 40 years of age or older
4. Smoking history of more than 10 pack years

Exclusion criteria:

1. Significant disease other than COPD
2. Clinically relevant abnormal lab values
3. History of asthma
4. Diagnosis of thyrotoxicosis
5. Diagnosis of paroxysmal tachycardia
6. A marked baseline prolongation of QT/QTc interval
7. A history of additional risk factors for Torsade de Pointes (TdP)
8. History of myocardial infarction within 1 year of screening visit
9. Unstable or life-threatening cardiac arrhythmia
10. Hospitalization for heart failure within the past year
11. Known active tuberculosis
12. Malignancy for which patient has undergone resection, radiation therapy or chemotherapy within last five years
13. History of life-threatening pulmonary obstruction
14. History of cystic fibrosis
15. Clinically evident bronchiectasis
16. History of significant alcohol or drug abuse
17. Thoracotomy with pulmonary resection
18. Oral ß-adrenergics
19. Oral corticosteroid medication at unstable doses
20. Regular use of daytime oxygen therapy for more than one hour per day
21. Pulmonary rehabilitation program in the six weeks prior to the screening visit
22. Investigational drug within one month or six half lives (whichever is greater) prior to screening visit
23. Known hypersensitivity to ß-adrenergic drugs, anticholinergics, BAC, EDTA
24. Pregnant or nursing women
25. Women of childbearing potential not using a highly effective method of birth control
26. Patients who have previously been randomized in this study or are currently participating in another study
27. Patients who are unable to comply with pulmonary medication restrictions
28. Patients with narrow-angle glaucoma or micturition disorder due to prostatic hyperplasia etc
29. Patients being treated with medications that prolong the QT/QTc interval

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2012-10; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 1237.24.24001 Boehringer Ingelheim Investigational Site, Toshima-ku, Tokyo, Japan

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This is a randomised, open-label, parallel group trial in which 3 weeks of randomised treatment are preceded by 2-week screening period and followed by 3-week follow-up period.
Groups:
- Tiotropium + Olodaterol (5µg/5µg): Oral inhalation of tiotropium 5 microgram (µg) (high dose) + olodaterol solution 5µg fixed-dose combination (FDC). The patients inhale 2 puffs from the RESPIMAT inhaler, once a day, in the morning up to 3 weeks.
- Tiotropium + Olodaterol (2.5µg/5µg): Oral inhalation of tiotropium 2.5 microgram (µg) (low dose) + olodaterol solution 5µg fixed-dose combination (FDC). The patients inhale 2 puffs from the RESPIMAT inhaler, once a day, in the morning up to 3 weeks.
Period: Overall Study
Arm/Group | Tiotropium + Olodaterol (5µg/5µg) | Tiotropium + Olodaterol (2.5µg/5µg)
Started | 16 (started are actually the randomized) | 16 (started are actually the randomized)
Completed | 13 | 16
Not Completed | 3 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Protocol Violation | 1 | 0
Not completed — other than stated above | 1 | 0

BASELINE CHARACTERISTICS:
Population: Treated Set (TS) includes all randomised patients who received at least one dose of trial medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | Tiotropium + Olodaterol (5µg/5µg) | Tiotropium + Olodaterol (2.5µg/5µg) | Total
Number analyzed (Participants) | 16 | 16 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.4 (10.5) | 69.4 (7.8) | 66.4 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 16 | 16 | 32

OUTCOME MEASURES:

1. Primary Outcome: Cmax,ss (Olodaterol)
Description: Maximum measured concentration of olodaterol after multiple inhaled administration of tiotropium+olodaterol in plasma at steady state (Cmax,ss).
  Per Protocol there are no primary endpoints defined. Therefore this pharmacokinetic endpoint was selected for primary outcome measure type.
Time Frame: 15 minutes (min) pre-dose and 5, 10, 20, 40 min, 1, 2, 3, and 4 hours (h) following drug administration on day 21
Population: The Pharmacokinetic (PK) set was defined as all treated patients who have at least 1 PK parameter in the treatment period without PK related important protocol violations. Two patients prematurely stopped the trial medication and had no PK measurement at Visit 3 (day 21) and were excluded from the PK set. Thus, the PK set included 30 patients.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: picogram/milliliter (pg/mL)
Arm/Group | Tiotropium + Olodaterol (5µg/5µg) | Tiotropium + Olodaterol (2.5µg/5µg)
Number analyzed (Participants) | 13 | 15
picogram/milliliter (pg/mL) | 4.33 (53.7) | 2.82 (106)

2. Primary Outcome: AUCt1-t2,ss (Olodaterol)
Description: Area under the concentration-time curve of olodaterol in plasma after multiple inhaled administration of tiotropium+olodaterol over the time interval 0 to 4 hours at steady state (AUCt1-t2,ss).
  Per Protocol there are no primary endpoints defined. Therefore this pharmacokinetic endpoint was selected for primary outcome measure type.
Time Frame: 15 min pre-dose and 5, 10, 20, 40 min, 1, 2, 3, and 4 h following drug administration on day 21
Population: The Pharmacokinetic (PK) set.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg*h/mL
Arm/Group | Tiotropium + Olodaterol (5µg/5µg) | Tiotropium + Olodaterol (2.5µg/5µg)
Number analyzed (Participants) | 12 | 13
pg*h/mL | 9.94 (29.9) | 8.14 (65.5)

3. Primary Outcome: AUC0-tz,ss (Olodaterol)
Description: Area under the concentration-time curve of olodaterol after multiple inhaled administration of tiotropium+olodaterol in plasma over the time interval from 0 to the time of the last quantifiable data point at steady state (AUC0-tz,ss).
  Per Protocol there are no primary endpoints defined. Therefore this pharmacokinetic endpoint was selected for primary outcome measure type.
Time Frame: 15 min pre-dose and 5, 10, 20, 40 min, 1, 2, 3, and 4 h following drug administration on day 21
Population: The Pharmacokinetic (PK) set.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg*h/mL
Arm/Group | Tiotropium + Olodaterol (5µg/5µg) | Tiotropium + Olodaterol (2.5µg/5µg)
Number analyzed (Participants) | 12 | 14
pg*h/mL | 9.94 (29.9) | 6.85 (105)

4. Primary Outcome: Tmax,ss (Olodaterol)
Description: Time from dosing to the maximum concentration of Olodaterol after multiple inhaled administration of tiotropium+olodaterol in plasma at steady state (tmax,ss).
  Per Protocol there are no primary endpoints defined. Therefore this pharmacokinetic endpoint was selected for primary outcome measure type.
Time Frame: 15 min pre-dose and 5, 10, 20, 40 min, 1, 2, 3 and 4 hours (h) following drug administration on day 21
Population: The Pharmacokinetic (PK) set.
Measure: Median (Full Range); unit: h
Arm/Group | Tiotropium + Olodaterol (5µg/5µg) | Tiotropium + Olodaterol (2.5µg/5µg)
Number analyzed (Participants) | 13 | 15
h | 0.183 [0.100 to 0.333] | 0.217 [0.100 to 2.00]

5. Primary Outcome: Aet1-t2,ss (Olodaterol)
Description: Amount of olodaterol that is eliminated in urine after multiple inhaled administration of tiotropium+olodaterol over the time interval 0 to 4 hours at steady state (Aet1-t2,ss).
  Per Protocol there are no primary endpoints defined. Therefore this pharmacokinetic endpoint was selected for primary outcome measure type.
Time Frame: from 0 to 4 hours following drug administration on day 21
Population: The Pharmacokinetic (PK) set.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram (ng)
Arm/Group | Tiotropium + Olodaterol (5µg/5µg) | Tiotropium + Olodaterol (2.5µg/5µg)
Number analyzed (Participants) | 13 | 16
nanogram (ng) | 74.8 (100) | 50.0 (123)

6. Primary Outcome: fe t1-t2,ss (Olodaterol)
Description: Fraction eliminated in urine from the time point t1 (0 h) to time point t2 (4 h) at steady state (fet1-t2,ss).
  Per Protocol there are no primary endpoints defined. Therefore this pharmacokinetic endpoint was selected for primary outcome measure type.
Time Frame: from 0 to 4 hours following drug administration on day 21
Population: The Pharmacokinetic (PK) set.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: percentage of dose
Arm/Group | Tiotropium + Olodaterol (5µg/5µg) | Tiotropium + Olodaterol (2.5µg/5µg)
Number analyzed (Participants) | 13 | 16
percentage of dose | 1.50 (100) | 0.999 (123)

7. Primary Outcome: CLR,t1-t2,ss (Olodaterol)
Description: Renal clearance from the time point t1 (0 h) until the time point t2 (4 h) at steady state (CLR,t1-t2,ss).
  Per Protocol there are no primary endpoints defined. Therefore this pharmacokinetic endpoint was selected for primary outcome measure type.
Time Frame: from 0 to 4 hours following drug administration on day 21
Population: The Pharmacokinetic (PK) set.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/min
Arm/Group | Tiotropium + Olodaterol (5µg/5µg) | Tiotropium + Olodaterol (2.5µg/5µg)
Number analyzed (Participants) | 12 | 13
mL/min | 152 (48.7) | 148 (42.8)

8. Secondary Outcome: Number of Participants With Adverse Events (Including Assessment Based on Physical Examination)
Description: Outcome data show are the number of patients with an adverse event including the assessment based on physical examination.
Time Frame: up to 6 weeks (3 weeks treatment and 3 weeks follow-up) post dose
Population: Treated Set (TS) includes all randomised patients who received at least one dose of trial medication.
Measure: Number; unit: participants
Groups:
- Tiotropium + Olodaterol (5µg/5µg): Oral inhalation of tiotropium 5 microgram (µg) (high dose) + olodaterol solution 5µg fixed-dose combination (FDC).The patients inhale 2 puffs from the RESPIMAT inhaler, once a day, in the morning up to 3 weeks.
- Tiotropium + Olodaterol (2.5µg/5µg): Oral inhalation of tiotropium 2.5 microgram (µg) (low dose) + olodaterol solution 5µg fixed-dose combination (FDC).The patients inhale 2 puffs from the RESPIMAT inhaler, once a day, in the morning up to 3 weeks.
Arm/Group | Tiotropium + Olodaterol (5µg/5µg) | Tiotropium + Olodaterol (2.5µg/5µg)
Number analyzed (Participants) | 16 | 16
participants | 4 | 2

9. Primary Outcome: Cmax,ss (Tiotropium)
Description: Maximum measured concentration of tiotropium after multiple inhaled administration of tiotropium+olodaterol in plasma at steady state (Cmax,ss).
  Per Protocol there are no primary endpoints defined. Therefore this pharmacokinetic endpoint was selected for primary outcome measure type.
Time Frame: 15 minutes (min) pre-dose and 5, 10, 20, 40 min, 1, 2, 3, and 4 hours (h) following drug administration on day 21
Population: The Pharmacokinetic (PK) set.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: picogram/milliliter (pg/mL)
Arm/Group | Tiotropium + Olodaterol (5µg/5µg) | Tiotropium + Olodaterol (2.5µg/5µg)
Number analyzed (Participants) | 13 | 14
picogram/milliliter (pg/mL) | 16.5 (92.0) | 6.49 (50.4)

10. Primary Outcome: AUCt1-t2,ss (Tiotropium)
Description: Area under the concentration-time curve of tiotropium in plasma after multiple inhaled administration of tiotropium+olodaterol over the time interval 0 to 2 hours at steady state (AUCt1-t2,ss).
  Per Protocol there are no primary endpoints defined. Therefore this pharmacokinetic endpoint was selected for primary outcome measure type.
Time Frame: 15 min pre-dose and 5, 10, 20, 40 min, 1 and 2 h following drug administration on day 21
Population: The Pharmacokinetic (PK) set.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg*h/mL
Arm/Group | Tiotropium + Olodaterol (5µg/5µg) | Tiotropium + Olodaterol (2.5µg/5µg)
Number analyzed (Participants) | 12 | 11
pg*h/mL | 14.8 (50.7) | 7.00 (52.8)

11. Primary Outcome: AUC0-tz,ss (Tiotropium)
Description: Area under the concentration-time curve of tiotropium after multiple inhaled administration of tiotropium+olodaterol in plasma over the time interval from 0 to the time of the last quantifiable data point at steady state (AUC0-tz,ss).
  Per Protocol there are no primary endpoints defined. Therefore this pharmacokinetic endpoint was selected for primary outcome measure type.
Time Frame: 15 min pre-dose and 5, 10, 20, 40 min, 1, 2, 3, and 4 h following drug administration on day 21
Population: The Pharmacokinetic (PK) set.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg*h/mL
Arm/Group | Tiotropium + Olodaterol (5µg/5µg) | Tiotropium + Olodaterol (2.5µg/5µg)
Number analyzed (Participants) | 12 | 13
pg*h/mL | 23.3 (44.8) | 7.99 (131)

12. Primary Outcome: Tmax,ss (Tiotropium)
Description: Time from dosing to the maximum concentration of tiotropium after multiple inhaled administration of tiotropium+olodaterol in plasma at steady state (tmax,ss).
  Per Protocol there are no primary endpoints defined. Therefore this pharmacokinetic endpoint was selected for primary outcome measure type.
Time Frame: 15 min pre-dose and 5, 10, 20, 40 min, 1, 2, 3, 4 hours following drug administration on day 21
Population: The Pharmacokinetic (PK) set.
Measure: Median (Full Range); unit: h
Arm/Group | Tiotropium + Olodaterol (5µg/5µg) | Tiotropium + Olodaterol (2.5µg/5µg)
Number analyzed (Participants) | 13 | 14
h | 0.100 [0.100 to 0.333] | 0.100 [0.083 to 0.183]

13. Primary Outcome: Aet1-t2,ss (Tiotropium)
Description: Amount of tiotropium that is eliminated in urine after multiple inhaled administration of tiotropium+olodaterol over the time interval 0 to 4 hours at steady state (Aet1-t2,ss).
  Per Protocol there are no primary endpoints defined. Therefore this pharmacokinetic endpoint was selected for primary outcome measure type.
Time Frame: from 0 to 4 hours following drug administration on day 21
Population: The Pharmacokinetic (PK) set.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram (ng)
Arm/Group | Tiotropium + Olodaterol (5µg/5µg) | Tiotropium + Olodaterol (2.5µg/5µg)
Number analyzed (Participants) | 13 | 16
nanogram (ng) | 336 (119) | 122 (118)

14. Primary Outcome: fe t1-t2,ss (Tiotropium)
Description: as for outcome 6
Time Frame: from 0 to 4 hours following drug administration on day 21
Population: The Pharmacokinetic (PK) set.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: percentage of dose
Arm/Group | Tiotropium + Olodaterol (5µg/5µg) | Tiotropium + Olodaterol (2.5µg/5µg)
Number analyzed (Participants) | 13 | 16
percentage of dose | 6.72 (119) | 4.89 (118)

15. Primary Outcome: CLR,t1-t2,ss (Tiotropium)
Description: Renal clearance from the time point t1 (0 h) until the time point t2 (4 h) at steady state (CLR,t1-t2,ss).
  Per Protocol there are no primary endpoints defined. Therefore this pharmacokinetic endpoint was selected for primary outcome measure type.
  Plasma concentration of tiotropium could not be quantified up to 4 hours for Tiotropium + Olodaterol (2.5μg/5μg).
Time Frame: from 0 to 4 hours following drug administration on day 21
Population: The Pharmacokinetic (PK) set.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/min
Arm/Group | Tiotropium + Olodaterol (5µg/5µg)
Number analyzed (Participants) | 12
mL/min | 292 (44.6)

16. Secondary Outcome: Number of Participants With Clinically Relevant Abnormalities in Vital Signs, Clinical Laboratory Tests and ECG
Description: Outcome data show are the number of participants with clinically relevant abnormalities reported as an adverse event (AE) related to the vital signs (pulse rate and blood pressure in supine position), clinical laboratory (routine blood chemistry, haematology, and urinalysis) tests and ECG (12-lead holter monitoring Electrocardiography). Relevant findings or worsening of baseline conditions were reported as adverse events.
  There were no clinically relevant abnormalities reported as an AE related to the vital signs and ECG.
Time Frame: up to 6 weeks (3 weeks treatment and 3 weeks follow-up) post dose
Population: The treated Set (TS).
Measure: Number; unit: participants
Arm/Group | Tiotropium + Olodaterol (5µg/5µg) | Tiotropium + Olodaterol (2.5µg/5µg)
Number analyzed (Participants) | 16 | 16
participants
  AEs reported related to vital signs | 0 | 0
  AEs reported related to ECG | 0 | 0
  Haematuria | 0 | 1
  Blood creatine phosphokinase increased | 1 | 0
  Blood urine present | 1 | 0

ADVERSE EVENTS:
Time Frame: up to 44 days (23 days maximum number of days a study treatment was used after first intake and 21 days follow-up)
Arm/Group | Tiotropium + Olodaterol (5µg/5µg) | Tiotropium + Olodaterol (2.5µg/5µg)
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 4/16 | 2/16
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tiotropium + Olodaterol (5µg/5µg) (N=16) | Tiotropium + Olodaterol (2.5µg/5µg) (N=16)
Bronchitis (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 1
Blood creatine phosphokinase increased (Investigations) | 1 | 0
Blood urine present (Investigations) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.